CLINICAL TRIAL: NCT06110533
Title: Descriptive Epidemiological Study of Hospitalized Children for Pulmonary Tuberculosis at Strasbourg University Hospitals
Brief Title: Epidemiological Study of Hospitalized Children for Pulmonary Tuberculosis at Strasbourg University Hospitals
Acronym: TPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8907
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary tuberculosis; Tuberculosis in children; Childhood tuberculosis; Mycobacterium tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary tuberculosis is the most common form of tuberculosis in children; According to the WHO, tuberculosis pulmonary tuberculosis in children represents approximately 80% of all cases of tuberculosis in children. In 2020, there were approximately 1.0 million new cases of pulmonary tuberculosis among children worldwide.

In France, childhood tuberculosis remains a rare disease; the most recent data show a rate of 3.3 cases per 100,000 inhabitants among children under 15 years old in 2019.

Pulmonary tuberculosis in children can lead to complications such as bronchiectasis and pneumothorax. Children living in homes where an adult has a active tuberculosis, or children with diseases chronic, malnourished or suffering from HIV are more likely to contract tuberculosis.

The aim of this research is to determine the incidence, identify the risk factors as well as the clinical forms of pulmonary tuberculosis in children hospitalized at Strasbourg University Hospitals between 2012 and 2022.

ELIGIBILITY:
Inclusion Criteria:

* Child (1 to 17 years old)
* Child hospitalized for pulmonary tuberculosis at Strasbourg University Hospital between January 1, 2012 and December 31, 2022.
* Child and/or his/her parental authority who have not expressed their opposition to the reuse of data for scientific research purposes.

Exclusion Criteria:

- Subject and/or their parental authority having expressed their opposition to the re-use of the child's data for scientific research purposes.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child (1 to 17 years old) hospitalized for pulmonary tuberculosis at Strasbourg University Hospital between January 1, 2012 and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04-14 (Estimated)

PRIMARY OUTCOMES:
Incidence and risk factors for pulmonary tuberculosis in children hospitalized at Strasbourg University Hospital between 2012 and 2022 | 1 month after hospitalization for pulmonary tuberculosis

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Ressources et de Compétences de la Mucoviscidose (CRCM) - CHU de Strasbourg - France, Strasbourg, France